CLINICAL TRIAL: NCT05896709
Title: A Novel Integrative Non-invasive Embryo Selection Approach for in Vitro Fertilization Based on Artificial Intelligence Enhanced Morphokinetic Analysis and Raman Spectra in Spent Culture Media
Brief Title: A Novel Integrative Non-invasive Embryo Selection Approach for IVF Based on MK-RS Analysis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Chung Pui Wah Jacqueline, Associate Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2022.661
Record Dates: First submitted 2023-05-10; First posted 2023-06-09 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Reproductive Issues; Subfertility; IVF
Keywords: non-invasive; in vitro fertilization; time-lapse imaging; artificial intelligence; morphokinetic analysis; Raman spectroscopy; embryo selection
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MK-RS (Experimental): Patients' embryos will be selected by MK-RS integrative analytical method.
  Interventions: Other: MK-RS
- Conventional (No Intervention): Patients' embryos will be selected by conventional method (i.e by embryologists).

INTERVENTIONS:
Other: MK-RS — The embryos are assessed by the AI-enhanced MK analysis together with RS analysis.
  Arms: MK-RS

SUMMARY:
During assisted reproductive technology treatment, embryo selection is an important process that may affect the clinical pregnancy rate. Many assisted reproductive technology units over the world have tried different approaches to increase the clinical pregnancy rate. Conventionally, the morphology of the embryo is assessed by the embryologist with naked eyes only. Nowadays, artificial intelligence (AI) has been used to assist in morphological assessment of the embryo. Our pilot study showed that the AI-enhanced morphokinetic (MK) analysis increased the accuracy in embryo selection by ~9%, while the detection rate for abnormal chromosomes in embryo has also been increased by Raman spectroscopy (RS) analysis. The combined MK-RS analysis will be able to complete embryo assessment within 5-6 days after fertilization. This method needs shorter time and is at lower cost when compared to invasive preimplantation genetic testing for aneuploidies (PGT-A).

In this study, we have combined the following non-invasive techniques to assist in embryo screening.

1. Using time-lapse imaging (i.e. images of embryo being taken every 10 minutes inside the incubator) with AI)-enhanced MK analysis to assess the entire morphological changes of the embryo.
2. As the embryo releases metabolites during its growth, the spent culture medium will be collected after culture of the embryo and then be used for RS analysis, which is a kind of metabolomics-based non-invasive PGT-A, for screening chromosomal abnormalities of the embryo.

This study will include two phases. In Phase I, it is a retrospective part. We will collect data to train the convolutional neural network (CNN)-enhanced MK with RS method on embryo selection, leading to the integrated approach (MK-RS). In Phase II, it is a randomized controlled trial and participants will be randomised into 2 groups. For the experimental group, embryo selection will be based on the MK-RS method, whereas embryo selection for the control group will rely on the traditional embryo assessment results alone. Then we will assess the clinical pregnancy rate and evaluate the efficacy of our approach finally. Patients who receive in vitro fertilisation (IVF)/ intracytoplasmic sperm injection (ICSI) treatment from The Assisted Reproductive Technology (ART) Unit of The Chinese University of Hong Kong, Prince of Wales Hospital will be recruited.

DETAILED DESCRIPTION:
Our study will include two phases. In Phase I (a retrospective study), archived data will be collected to train the CNN-enhanced MK with RS method on embryo selection, leading to the integrated approach (MK-RS). In Phase II (a prospective study), the integrated MK-RS method established will be used to select embryos, assess the clinical pregnancy rate and evaluate the efficacy of our approach in a randomized controlled trial.

In Phase I, images of the embryo will be captured every 10 minutes by the in-built microscope and camera in the time-lapse incubator. Images will then be assessed by the CNN algorithm for day one human embryo segmentation to identify three distinct features: the zona pellucida (ZP), cytoplasm and pronucleus (PN). The morphodynamics of these three features during the fertilisation to first division will be wrapped up as time series data for the integration. The morphology changes after the first division will be semi-auto annotated, which will be analysed by the commercial MK scoring system (KID Score).

After removal of embryos/blastocysts from the culture dish, the corresponding spent culture medium (SCM) will be collected in sterile polymerase chain reaction (PCR) tubes. Blank culture mediums will also be collected with the same operating standard. A specifically designed sampler will be used to pipette 7μL SCM of each sample, passing through the oil layer of the SCM, and then drop it onto a disposable quartz glass slide and illuminated by RS system (Basecare Raman 200, China). The RS system will be calibrated to 520.5 cm-1 by silicon wafer before testing. Laser excitation parameters are set as follows: 785 nm wavelength, 320 mW power and 100 μm laser spot diameter. Signals are captured in standard mode with a chargecoupled device (CCD) camera with a 20-seconds integration time. Three replicates will be done for each aliquot. Re-calibration is essential when different culture media is tested, considering that G-1 medium is used for embryos before Day 3 and G-2 medium is used for embryos after Day 3. All obtained spectra will be pre-processed by subtracting the background signal. Spectroscopy signals within the near-infrared region (600 cm-1- 1800 cm-1) are analysed for vector normalisation using Labspec 6 software (Horiba, Japan). Our previous SCM samples with known TE ploidy results will be used as a training dataset to establish euploid-aneuploid classification standards. Stacking classification algorithm will be adopted, considering its high overall accuracy (95.9%, unpublished data).

As the segmented time series of CNN algorithm, KID Score annotations and RS profiling results have hundreds of subparameters, we will assemble them together with the ensemble learning, which considers each subparameter as a weak classifier and re-allocated their weights during the training. The primary index for the training is the clinical pregnancy outcome and for the ultimation of the information beneath CNN-enhanced MK and RS, the blastocyst formation results will be used as a secondary index. The ratio of the training set and test set will be 1:1 and in the training set, a 5-fold cross-validation will be performed for monitoring the overfitting.

Phase II will comprise a prospective, single-blinded, randomised controlled trial designed to validate the trained MK-RS method for embryo selection. Metabolomic SCM profiling using RS with CNN-enhanced MK analysis will be used to assess embryo developmental potential along with traditional morphological embryo assessments. The embryo developmental potential results will be used to select the best quality of embryos. Sensitivity and specificity will be assessed using the patient's TE biopsy or non-invasive prenatal testing (NIPT) results will further confirm the scoring of MK-RS method, if available.

Randomisation:

In Phase II, participants who fulfil all the inclusion and exclusion criteria and consent to join the study will be randomised into experimental group and control group in 1 to 1 ratio using a computer-generated randomisation list. For the experimental group, embryo selection will be based on the MK-RS method established in Phase I, whereas embryo selection for the control group will rely on the traditional embryo morphology grading results alone. All participants will be blinded in this trial.

ELIGIBILITY:
Inclusion Criteria:

1. Patients undergoing IVF/ ICSI treatment
2. Patients receiving the first, second or third IVF/ICSI treatment cycle
3. Patients and their partners willing to sign the informed consent agreement
4. Patients having at least three normal fertilised embryos on the day of the fertilization check
5. Consecutive women undergoing IVF treatment
6. Patients planning to use a time-lapse incubator for embryo culture

Exclusion Criteria:

1. Day one human embryos with blur imaging
2. Large obstructions in the embryo area
3. More than half of the embryo area is blocked by the well or degeneration
4. Patients with more than half of the embryos without sufficient spent culture medium for RS analysis
5. Patients with known genetic diseases

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 176 (Estimated)
Dates: Start 2023-07-17 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Clinical pregnancy rate | 6-8 weeks of gestation
  To assess for the presence of gestational sac using ultrasonography after embryo transfer procedure

SECONDARY OUTCOMES:
Miscarriage rate | 4-24 weeks of gestation of the participants
  To assess for any miscarriage if participants get pregnant after embryo transfer procedure
Multiple pregnancy rate | 6-8 weeks of gestation
  To assess for the presence of two or more gestational sacs using ultrasonography after embryo transfer procedure
Ploidy status | Within 10 days after the embryos are fertilised, or 4-40 weeks of gestation
  To assess the ploidy status of the embryo for patients who have underwent non-invasive prenatal testing (NIPT) or genetic testing during ART treatment or antenatal care
Live birth rate | From 24 weeks of gestation up to 40 weeks
  To assess whether live babies are born after ART treatment

CONTACTS AND LOCATIONS:
Overall Officials: PUI WAH JACQUELINE CHUNG, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- The Chinese University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No